CLINICAL TRIAL: NCT05576584
Title: Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Food Effects of GST-HG121 Tablets in Single and Multiple Administration in Chinese Adult Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetic Characteristics Evaluation on GST-HG121 Tablets
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Akeylink Biotechnology Co., Ltd. (Industry)
Collaborators: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: GST-HG121-I-01
Record Dates: First submitted 2022-08-31; First posted 2022-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-07

CONDITIONS: Pharmacokinetics; Food Affect; Single Ascending Dose; Maximum Applicable Dose
Keywords: Pharmacokinetics; food affects; Single Ascending Dose; Maximum Applicable Dose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose (Placebo Comparator): Five dose groups: 5mg (group I), 15mg (Group II), 30mg (Group III), 60mg (Group IV) and 100mg (Group V). According to the safety, tolerance and PK parameters of group V, higher dose group studies (150mg and 200mg alternatively) are not excluded. There were 10 subjects in each group, of which 8 received GST-HG121 tablets and 2 received placebo.
  Interventions: Drug: GST-HG121 tablets; Drug: Placebo
- Multiple Ascending Dose (Placebo Comparator): According to the results of single dose study, it is planned to select 1-3 dose groups within the range of single dose for oral administration for 7 consecutive days. There were 12 subjects in each group, of which 10 received GST-HG121 tablets and 2 received placebo. From D 1 to d 7, take GST-HG121 tablets or placebo orally on an empty stomach every day, tentatively once a day (the specific administration frequency may be adjusted based on the results of the single dose increase test)
  Interventions: Drug: GST-HG121 tablets; Drug: Placebo
- food affects（A） (Placebo Comparator): 10 subjects (8 received GST-HG121 tablets and 2 received placebo)
  Interventions: Drug: GST-HG121 tablets; Drug: Placebo
- food affects（B） (Active Comparator): 8 subjects (all received GST-HG121 tablets)
  Interventions: Drug: GST-HG121 tablets; Drug: Placebo

INTERVENTIONS:
Drug: GST-HG121 tablets — This trial includes single-dose studies and multiple-dose studies, The single-dose study included 5 dose groups of 5 mg, 15 mg, 30 mg, 60 mg, 100 mg（Alternative groups include 150mg and 200mg）. Based on the results of a single dose, select 1 to 3 doses which are tolerated in SAD to conduct multiple dose studies.
Drug: Placebo — This trial includes single-dose studies and multiple-dose studies, The single-dose study included 5 dose groups of 5 mg, 15 mg, 30 mg, 60 mg, 100 mg（Alternative groups include 150mg and 200mg）. Based on the results of a single dose, select 1 to 3 doses which are tolerated in SAD to conduct multiple dose studies.

SUMMARY:
This phase I clinical study is a phase I clinical study on the safety, tolerability, pharmacokinetic characteristics and food effects of single / continuous administration in Chinese adult healthy subjects

DETAILED DESCRIPTION:
This study will be divided into three parts: single dose escalation (SAD) study, multiple dose escalation (MAD) study and food impact study. The sad study and mad study adopted a randomized, double-blind, placebo-controlled, dose increasing trial design to evaluate the safety, tolerability and pharmacokinetic characteristics of gst-hg121 tablets. A randomized, two cycle, double crossover trial design was adopted for the study of food effects. Healthy Chinese adult volunteers were randomly divided into two groups. In the first cycle, the drug was administered on an empty stomach and after a meal, and in the second cycle, the drug was administered on an empty stomach and after a meal to evaluate the effects of food on the pharmacokinetic characteristics of gst-hg121 tablets.

Part I: Study on single dose increment A total of 5 dose groups were set for a single administration: 5mg (group I), 15mg (Group II), 30mg (Group III), 60mg (Group IV) and 100mg (Group V). According to the safety, tolerance and PK parameters of group V, higher dose group studies (150mg and 200mg are not excluded). There were 10 subjects in each group, of which 8 received gst-hg121 tablets and 2 received placebo. Therefore, it is planned to recruit 50 subjects to study the safety, tolerance and pharmacokinetics of single administration. Each group was administered once, and gst-hg121 tablet or placebo was orally administered once under the fasting condition of D1. The subjects will be kept in the hospital to observe the vital signs and whether there are adverse events. Safety inspection is required at D2, D4 and D6, tolerance evaluation is required at D6, and pharmacokinetic indexes of gst-hg121 are detected at the same time.

Subjects in different dose groups will be enrolled in the group in turn. After all the subjects in one group have completed the evaluation, the researchers and the sponsor will jointly evaluate the safety, tolerance and PK parameters under the dose level to determine whether to conduct the next dose group study. If necessary, relevant clinical experts can be invited to consult and make decisions. After obtaining the PK report of the first dose group, it is possible to adjust the time point of collection or inspection of PK samples or other inspection items. After the completion of all 5 dose groups, the single dose increment test will be terminated. If the tolerance and safety of the drug at the highest dose are good, the investigator and the sponsor shall conduct a comprehensive evaluation, and it is not excluded to conduct the trial of the higher dose standby group (> 100mg).

Part II: Study on multiple dose escalation According to the results of single dose study, it is planned to select 1-3 dose groups within the range of single dose for oral administration test for 7 consecutive days (the specific dose group is determined according to the results of single dose increment test). There were 12 subjects in each group, of which 10 received gst-hg121 tablets and 2 received placebo. Therefore, it is planned to recruit 36 subjects for safety, tolerance and pharmacokinetics study of multiple administration. From D 1 to d 7, take gst-hg121 tablets or placebo orally on an empty stomach once a day (the specific administration frequency may be adjusted based on the results of the single dose increment test). After the first administration, conduct safety inspection on D3, D6 and D12, and conduct tolerance evaluation on D12.

After a group of subjects have completed the evaluation, the researcher and the sponsor will jointly evaluate the safety, tolerance and PK parameters at the dose level to determine whether to conduct the next dose group study. If necessary, relevant clinical experts can be invited to consult and make decisions. After obtaining the PK results of the first dose group in the multiple dose increment test, it is possible to adjust the time point of collection or inspection of PK samples or other inspection items. After the multiple dose increasing test is terminated, the investigator and the sponsor shall conduct comprehensive evaluation, and it is not excluded to select other doses within the safe dose range for further test.

Part III: Food impact study The 30mg (Group III) dose group or 60mg (Group IV) dose group (the final dose is determined according to the results of the single dose study) is tentatively determined, and the single dose, food impact and drug metabolism and transformation studies need to be completed. 18 subjects are planned to be enrolled into the group and divided into two groups: 10 subjects in group A (including 8 subjects receiving gst-hg121 tablets and 2 subjects receiving placebo) and 8 subjects in group B (all receiving gst-hg121 tablets). Subjects in group a need to participate in the study on the effects of single administration of 30mg or 60mg and food on pharmacokinetics, and subjects in group B need to participate in the study on the effects of food on pharmacokinetics and drug metabolism and transformation.

In group A, the first cycle was administered under the fasting condition of D1, and the second cycle was administered under the standard postprandial condition of one day of d8-d15. In group B, the first cycle was administered under the standard postprandial condition of D1, and the second cycle was administered under the fasting condition of one day of d8-d15. The two cycles were administered alternately, and the cleaning period was 7-14 days (the cleaning period was determined according to the results of the single administration study). The administration study of group A under fasting condition is equivalent to the single administration study of 30mg or 60mg gst-hg121 tablets. After the first administration, the safety inspection was conducted on D2, D4 and D6, and the tolerance evaluation was conducted on D6. If the first administration of group A is completed and the tolerance evaluation result indicates that it can be tolerated, the second cycle of group A and the first cycle of group B can be carried out.

During the trial, blood samples will be collected from the subjects at the time point planned in the protocol for pharmacokinetic analysis. As gst-hg121 tablet has not been applied in human body and there is no human PK parameter for reference, this study will be conducted by sentinel enrollment. Group I, group II, group III, group IV, group A and group V: two subjects were enrolled first (two subjects received the test drug gst-hg121 tablets, half male and half female), and the remaining eight subjects were enrolled after at least 48 hours of observation (the two subjects in the first group need to take blood samples and complete the drug concentration detection and data analysis. If it is necessary to fine tune the PK sample collection time point, it can be adjusted in group II). The fourth group (group B) included 8 subjects (all taking the test drug gst-hg121). Two subjects (taking the test drug gst-hg121 tablets, half male and half female) were enrolled in each dose group after multiple administration, and the remaining 10 subjects were enrolled in the group after at least 72 hours of observation.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects must give informed consent to the test before the test, fully understand the test content, process and possible adverse reactions, and voluntarily sign a written informed consent;
2. Able to complete the research according to the requirements of the test scheme;
3. Chinese male and female subjects aged between 18 and 55 years old (both inclusive).
4. The weight of male subjects shall not be less than 50kg and that of female subjects shall not be less than 45kg. Body mass index (BMI) = body weight (kg) / height 2 (M2), and the body mass index is within the range of 18-28 kg / m2 (including the critical value);
5. Effective contraceptive measures can be taken within 6 months from the start of screening to the last administration of the trial drug, and sperm and eggs donation shall be avoided during this period. See Appendix 5 for specific contraceptive measures;
6. At the time of screening, there was no history of respiratory, circulatory, digestive, urinary, blood, endocrine, nervous system diseases and metabolic abnormalities with clinical significance;
7. At the time of screening, the results of vital signs, physical examination, laboratory examination, electrocardiogram, abdominal color ultrasound (liver, gallbladder, spleen, pancreas, double kidneys) and chest X-ray (positive position) examination were normal or abnormal but judged by the investigator to have no clinical significance.

Exclusion Criteria:

1. Hospitalization within 30 days before the trial administration, or surgical operation within 6 months before the trial administration, or the presence of transplanted organs in the body, or any medical condition that is not suitable for participating in the trial according to the judgment of the investigator;
2. Those who have participated in other intervention clinical trials and used clinical study drugs within 3 months before the trial administration or plan to participate in other clinical studies at the same time during the study (if the subjects withdraw from the study before treatment, that is, they are not randomized or treated, they can be included in the study);
3. Have been vaccinated with live vaccine within 3 months before the trial administration, or need to be vaccinated during the study period;
4. Clinically significant drug allergy history or specific allergic disease history (asthma, urticaria) or known allergy to the test drug or its excipients;
5. Blood donation or massive blood loss (> 450 ml) or use of blood products or blood transfusion within three months before screening;
6. Those who smoked more than 5 cigarettes per day on average 3 months before the trial;
7. The subjects had a history of alcoholism within 12 months before the screening (drinking 14 units of alcohol every week: 1 unit = 285 ml of beer, 25 ml of liquor, or 100 ml of wine), or the subjects could not use any alcohol containing products within 72 hours before the test administration and during the whole test, or the subjects were positive in the alcohol breath test during the screening period;
8. Those with positive urine drug screening (morphine, marijuana) or drug abuse history;
9. Taking any prescription medicine, over-the-counter medicine, any health product or herbal medicine within 14 days before screening; Any drug that alters liver enzyme activity was taken 28 days before screening; Inhibitors or inducers combined with the following CYP3A4, P-gp or BCRP, such as itraconazole, ketoconazole or dronedarone;
10. Those who have taken special diet (including pitaya, mango, grapefruit, etc.) or had vigorous exercise or other factors affecting drug absorption, distribution, metabolism and excretion within 2 weeks before screening;
11. Recent major changes in diet or exercise habits;
12. Have a history of dysphagia or any gastrointestinal disease affecting drug absorption;
13. Suffering from any disease that increases the risk of bleeding, such as hemorrhoids, gastritis or gastric and duodenal ulcers;
14. Subjects who cannot tolerate standard meals (high-fat and high calorie meals) (this article is only applicable to subjects participating in food impact studies);
15. Female subjects are breastfeeding or preparing to become pregnant in the near future during the screening period or the test process, or the serum pregnancy results are positive;
16. Screening positive for hepatitis B surface antigen, hepatitis C antibody, AIDS antibody and Treponema pallidum antibody;
17. Ingestion of chocolate, any food or drink containing alcohol, caffeine or xanthine 24 hours before taking the study drug;
18. Subjects considered by the investigator to have other factors unsuitable for participating in the trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-12-28 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Treatment-Related Adverse Events | SAD up to Day 6 and MAD up to Day 12
  Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Area Under Curve (AUC) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
T1/2 | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Cl/F | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Ae(0~120h) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Fe(0~120h) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No